CLINICAL TRIAL: NCT07088224
Title: Analysis of Risk Factors and Establishment of Prediction Model for Postoperative Sore Throat After Thyroid Surgery Under General Anesthesia
Brief Title: Establishment of Prediction Model for Postoperative Sore Throat
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, XiaoLiang Wang, Chief Physician, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20250624-12
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Sore Throat
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational studies without intervention — Observational studies without intervention

SUMMARY:
This observational study aims to identify the risk factors associated with postoperative sore throat (POST) and to develop a clinical prediction model for patients undergoing thyroid surgery under general anesthesia. Despite improvements in surgical and anesthetic techniques, POST remains one of the most common complications following thyroidectomy, with an incidence of up to 80%. POST can significantly impact patient comfort, swallowing function, nutritional intake, and recovery quality, leading to prolonged hospitalization and increased healthcare costs.

The etiology of POST is multifactorial, involving intubation-related factors (e.g., endotracheal tube size, cuff pressure), surgery-related factors (e.g., duration of surgery, neck hyperextension), and patient-related factors (e.g., age, sex, smoking history, pre-existing throat symptoms). However, large-scale, systematic studies in the Chinese population remain limited.

With the increasing adoption of Enhanced Recovery After Surgery (ERAS) principles, the accurate identification of modifiable risk factors and early prediction of POST risk are essential for targeted preventive strategies and improved perioperative management. Recent advancements in machine learning and statistical modeling allow for the development of personalized, multifactorial risk assessment tools.

In this study, clinical data from patients undergoing thyroid surgery at Nanjing First Hospital will be collected and analyzed. The primary goal is to identify key preoperative and intraoperative predictors of POST and to establish a multivariable nomogram-based prediction model. Internal validation using bootstrap methods will be performed to evaluate the model's discrimination, calibration, and clinical utility, ultimately supporting evidence-based interventions to improve postoperative outcomes and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years； Undergoing thyroid surgery under general anesthesia, including both open and endoscopic procedures； Complete postoperative follow-up records available (minimum 48 hours)； Accessible and complete surgical and anesthesia records； Provision of written informed consent by the patient or their legally authorized representative；

Exclusion Criteria:

Failed tracheal intubation or need for emergency tracheotomy during surgery； Reoperation required due to postoperative complications such as bleeding or nerve injury； Severe cardiopulmonary disease (ASA physical status ≥ IV) or long-term use of corticosteroids； Incomplete clinical data；

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with postoperative thyroid surgery pain
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
incidence of Postoperative Sore rate within 24 hours after surgery | within 24 hours after surgery

SECONDARY OUTCOMES:
incidence of Postoperative Sore Throat rate 1 hour after surgery | 1 hour after surgery
incidence of Postoperative Sore Throat rate 48 hour after surgery | 48 hour after surgery